CLINICAL TRIAL: NCT00159445
Title: Phase II Study of Capecitabine and Gemcitabine in Patients With Metastatic Colorectal Cancer
Brief Title: Capecitabine and Gemcitabine in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3C-03-12
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Colorectal Cancer; Colon Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Gemcitabine; Capecitabine

INTERVENTIONS:
Drug: gemcitabine, capecitabine

SUMMARY:
This study is for patients with colorectal cancer that has spread and has increased in size after standard treatments. This study is being done to find out how long it takes their tumors to grow after treatment with the chemotherapy drugs capecitabine and gemcitabine. Capecitabine is a chemotherapy drug that has been approved by the FDA for the treatment of colorectal cancer. We are adding another drug (called gemcitabine), which is approved by the FDA for the treatment of cancer of the pancreas to see if the ability of capecitabine to shrink tumors can be improved by adding gemcitabine. The side effects of the combination will also be evaluated. Another purpose of this study is to measure the levels of certain substances that affect how the body reacts to the chemotherapy agents in cancer cells (in the tumor). In addition, the genes (which are the cell's blueprint for these substances) will also be evaluated in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic adenocarcinoma of the colon or rectum, with measurable disease. The primary histologic diagnosis is sufficient if there is clear evidence by imaging and/or markers of metastatic disease sites.
* Patients must have failed CPT-11 and oxaliplatin based therapies.
* Patients must have received at least two prior chemotherapy regimens for advanced disease (completed > 4 weeks prior to enrollment).
* Tumor must be accessible for biopsy or paraffin embedded tissue must be available for review.
* SWOG performance status 0-2.
* AGC >1000, platelets >100,000.
* Total bilirubin < 3 x upper limit of normal. Transaminase (AST and/or ALT) < 2 x upper limit of normal or < 5 x upper limit of normal in patients with liver metastasis.
* Patients must have a measured or calculated creatinine clearance greater than 35 mL/min obtained within 28 days prior to registration.
* Age greater than or equal to 18 years
* Patients should have hemoglobin > 9 g/dL; patients may be transfused to achieve this level of hemoglobin.
* Except for cancer-related abnormalities, patients should not have unstable or pre-existing major medical conditions.

Exclusion Criteria:

* History of a malignancy other than colon or rectal cancer, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for five years.
* Patients with brain metastasis.
* History of recent (within one year) myocardial infarction or evidence of congestive heart failure.
* Patients that have psychological, familial, sociological, or geographical conditions that do not permit medical follow-up and compliance with the study protocol.
* Patients should not have any immediate life-threatening complications of their malignancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2004-03; Primary Completion 2007-03 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To assess time to progression in patients with metastatic colorectal cancer treated with a combination of gemcitabine and capecitabine after progressing on two or more therapies for advanced disease, and having failed both CPT-11 and Oxaliplatin bas

SECONDARY OUTCOMES:
To assess the response rate and survival in patients with metastatic colorectal cancer treated with a combination of gemcitabine and capecitabine after progressing on two or more therapies for advanced disease. To assess the toxicity of this regimen.
To assess whether polymorphisms of thegenes involved in the 5-FU metabolic pathway are associated with efficacy of chemotherapy and toxicity.
To test the hypothesis that increased gene expression levels predict chemoresistance to capecitabine.

CONTACTS AND LOCATIONS:
Overall Officials: Syma Iqbal, M.D., Principal Investigator — U.S.C./Norris Comprehensive Cancer Center
Locations (1):
- U.S.C./Norris Comprehensive Cancer Center, Los Angeles, California, United States